CLINICAL TRIAL: NCT05820074
Title: Investigating Neural Biomarkers for Gait in Parkinson's Patients
Status: Recruiting | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: cereneo center for Neurology and Rehabilitation (Unknown); University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01382 NGB
Record Dates: First submitted 2022-12-13; First posted 2023-04-19 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: Parkinson's disease; gait parameters; neural activity; Percept PC; deep brain stimulation
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic | interventions — Electroencephalography; Motion Capture; Electromyography; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Young, healthy control: Young healthy participants below 45 years will take part in a gait protocol involving treadmill walking with pertubations and overground walking including obstacle stepping, figure-8-walk and timed-up-and-go test, as well as a seated-stepping section.
  During the protocol, neural activity is recorded using EEG.
  Interventions: Diagnostic Test: Neural Activity Recording; Diagnostic Test: Movement Parameter Recording
- Age-matched healthy control: Age-matched healthy participants above 45 years will take part in a gait protocol involving treadmill walking with pertubations and overground walking including obstacle stepping, figure-8-walk and timed-up-and-go test, as well as a seated-stepping section.
  During the protocol, neural activity is recorded using EEG.
  Interventions: Diagnostic Test: Neural Activity Recording; Diagnostic Test: Movement Parameter Recording
- Parkinson's patients: Parkinson's patients will take part in a gait protocol involving treadmill walking with pertubations and overground walking including obstacle stepping, figure-8-walk and timed-up-and-go test, as well as a seated-stepping section. Additionally, a neuromodulation set-up will be tested.
  During the protocol, neural activity is recorded using EEG and signals from the DBS-electrodes.
  Interventions: Diagnostic Test: Neural Activity Recording; Diagnostic Test: Movement Parameter Recording; Other: Neuromodulation

INTERVENTIONS:
Diagnostic Test: Neural Activity Recording — Neural Activity is measured using EEG in all groups. Additionally, in Parkinson's patients, local-field-potentials from deep brain stimulation electrodes are recorded.
  Other Names: Electroencephalography (EEG); Local-Field-Potentials with deep brain stimulation electrodes
Diagnostic Test: Movement Parameter Recording — Gait-related movement parameters are non-invasively recorded using motion capture, accelerometers and electromyography.
  Other Names: Motion capture; Accelerometers; Electromyography
Other: Neuromodulation — Neural signals are recorded with the electrodes of the deep brain stimulation device. Parkinson's patients are asked to modulate their neural activity by observing the streamed neural activity and applying mental strategies.
  Groups: Parkinson's patients

SUMMARY:
This observational study's main goal is to learn more about the neural mechanisms during movement in Parkinson's disease. Furthermore, it aims to inspire personalised treatment options.

Participants will undergo a protocol that involves walking and gait-related motor tasks, such as seated stepping. During the protocol, brain activity will be recorded.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is the second most common neurodegenerative disease accompanied by motor impairment [1]. Although symptomatic treatments like medication with Dopamine equivalents and deep brain stimulation (DBS) are available, the effects are very heterogeneous among patients and often cease over time.

This study aims to generate insights into the neural mechanisms of PD by determining neural biomarkers for gait. The insights of this study may further inspire personalised treatment approaches.

The primary objective is to identify neural biomarkers for gait. It is hypothesised that characteristic neural oscillations are underlying kinematic patterns in healthy participants and PD patients.

The secondary objective is to compare the neural activity during gait and a seated lower limb motor task between healthy participants and PD patients. To this end, the investigators hypothesise that neural correlates of gait and of a seated lower limb motor task differ between healthy participants and PD patients.

60 participants will be included, 30 healthy participants and 30 PD patients. All participants must be older than 18 years and give informed consent. Potential participants will be pre-screened and will be informed about the study via phone call/email. Before any study procedure, participants will give informed consent as documented by signature. Afterwards, inclusion/exclusion criteria, medical history and participant characteristics will be assessed. PD patients must be of postural instability and gait difficulty sub-type.

The study consists of one session of approximately 2.5 hours. During this session, electroencephalography (EEG) in healthy participants and EEG + local field potentials of the subthalamic nucleus from implanted DBS-electrodes in PD patients will be recorded during standardised gait sequences and a seated lower limb motor task. Furthermore, a short-term neuromodulation task will be investigated.

Gait-related parameters will be recorded using motion capture, surface electromyography (EMG) and accelerometers. Gait characteristics, including symmetry, coordination, variability, and resilience will be assessed. All recording devices are approved on the market. The protocol of the session slightly differs between healthy participants and PD patients since no DBS electrodes are implanted in healthy participants, but still allows for comparison between the groups.

ELIGIBILITY:
Inclusion Criteria:

All participants

* must have given informed consent as documented by signature
* agree to comply with the study procedures

Healthy control group

* no neurological, orthopedic, or rheumatologic disease history
* no identified sensory impairment.
* no epilepsy and self-diagnosed acute or chronic psychiatric disorders

Parkinson's Patients

* non-tremor dominant idiopathic PD patients
* presence of postural instability (UPDRS >1 for postural instability [17]), gait disturbance, and absence of other causes of reduced balance
* Implanted with Percept™ PC neurostimulator
* Able to be in the stimulation OFF

Exclusion Criteria:

* Relevant cognitive impairment, with a score on Montréal Cognitive Assessment (MoCA) < 20
* History of physical or neurological condition that interferes with study procedures
* Social and/or personal circumstances interfering with the ability to come to the session

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited among students, employees and associated persons of ETH Zürich, the University of Zürich, the University Hospital of Zürich, and Balgrist University Hospital and other centers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Cortical activity underlying kinematic gait patterns will be recorded by electroencephalograph of the healthy and Parkinson patients | 30 minutes
  Using a mobile EEG system to measure neural activity during walking
Electromyography (Delsys®) of the healthy and Parkinson patients | 30 minutes
  Electrodes will be attached to a representative lower limb muscle, such as the tibialis anterior.
Detect onset of task-related movements detected by an accelerometer that will be placed on the hand and foot of the healthy and the parkinson patients | 30 minutes
  ZurichMOVE® detects onset of movements

SECONDARY OUTCOMES:
Compare cortical activity between healthy subjects and parkinson patients | 30 minutes
  Neural activity between healthy controls and partient cohort will be compared.

OTHER OUTCOMES:
Difference in movement frequency between healthy participants and PD patients | 15 minutes
  Analysing the difference between healthy subjects and PD patients
Difference in the range of motion between healthy participants and PD patients | 15 minutes
  Analysing the difference between healthy subjects and PD patients

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lambercy, PhD, Principal Investigator — RELab, ETH Zürich
Locations (1):
- Cereneo, Vitznau, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Poewe W, Seppi K, Tanner CM, Halliday GM, Brundin P, Volkmann J, Schrag AE, Lang AE. Parkinson disease. Nat Rev Dis Primers. 2017 Mar 23;3:17013. doi: 10.1038/nrdp.2017.13. PMID 28332488
- [Background] Ravi DK, Gwerder M, Konig Ignasiak N, Baumann CR, Uhl M, van Dieen JH, Taylor WR, Singh NB. Revealing the optimal thresholds for movement performance: A systematic review and meta-analysis to benchmark pathological walking behaviour. Neurosci Biobehav Rev. 2020 Jan;108:24-33. doi: 10.1016/j.neubiorev.2019.10.008. Epub 2019 Oct 19. PMID 31639377
- [Background] Rodriguez-Oroz MC, Moro E, Krack P. Long-term outcomes of surgical therapies for Parkinson's disease. Mov Disord. 2012 Dec;27(14):1718-28. doi: 10.1002/mds.25214. Epub 2012 Dec 3. PMID 23208668
- [Background] Bichsel O, Stieglitz LH, Oertel MF, Baumann CR, Gassert R, Imbach LL. Deep brain electrical neurofeedback allows Parkinson patients to control pathological oscillations and quicken movements. Sci Rep. 2021 Apr 12;11(1):7973. doi: 10.1038/s41598-021-87031-2. PMID 33846456